CLINICAL TRIAL: NCT01140711
Title: Functional MRI Evaluation of Brain Response to Visual Food Stimulation in Morbidly Obese Patients Before and After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: SHEBA-7649-10-DG-CTIL
Record Dates: First submitted 2010-06-08; First posted 2010-06-09 (Estimated); Last update posted 2018-02-06 (Actual); Status verified 2018-02

CONDITIONS: Morbid Obesity; Satiety
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gastric bypass (Experimental): Patients submitted to gastric bypass for treatment of morbid obesity
  Interventions: Procedure: fMRI imaging following visual stimulation of food and non-food images
- Sleeve gastrectomy (Experimental): Patients submitted to sleeve gastrectomy for treatment of morbid obesity
  Interventions: Procedure: fMRI imaging following visual stimulation of food and non-food images

INTERVENTIONS:
Procedure: fMRI imaging following visual stimulation of food and non-food images — fMRI Scans will be performed in a 3 tesla MRI scanner. All subjects will be scanned for anatomical imaging without injection of contrast material. These structural images will be used to localize the functional data obtained. Functional test will include several measurements of brain activity while viewing visual stimuli.
  fMRI allows collection of information about brain activity with good spatial and temporal resolution. Protocols allow rapid assessment of regional activation in different brain regions during exposure to different visual stimuli.It provides a detailed functional map.
  Scan test protocol includes anatomical measurement - 3D FSPGE T1w sequence, Asset DTI and repeated fMRI measurements (based on echo EPI, T2 * w, BOLD sequences). Test paradigms include picture collections of various foods non-food objects similar in size, color and shape.

SUMMARY:
Aim of study:

To evaluate changes in feeding-related neural activity after different bariatric procedures in morbidly obese patients. Relationship of gut hormone levels will be assessed as well.

DETAILED DESCRIPTION:
Bariatric surgery mediates weight-loss via one or several mechanisms inherent to each technique used. Surgical restriction is the "lowest common denominator" shared, to various extent, by all procedures. Different degrees of malabsorption are utilized in "bypass procedures" such as Roux-Y gastric bypass (GBP), biliopancreatic diversion (BPD) and biliopancreatic diversion with duodenal switch (BPD-DS). These surgical options differ, also, in the degree of weight loss they promote. This difference is due to several factors including the extent of appetite suppression, increase in energy expenditure and degree of malabsorption achieved by the different procedures.

A post-operative change in the gut-brain hormonal axis is a component that has recently drawn much attention and research but is still ill defined. It is an effect, presumably mediated by a change in a myriad of peptides and hormones originating mostly from the intestinal tract, eliciting a change in hunger and satiety feelings as well as a change in the drive to eat. Generally speaking, patients after sleeve gastrectomy (SG) and the bypass procedures mentioned, have a decreased appetite and report a reduced drive to seek food, which presumably contributes to their weight loss.

Functional magnetic resonance imaging (fMRI) is an imaging modality which measures the hemodynamic response (change in blood flow) related to neural activity in the brain, therefore allowing mapping of areas in the brain which become active due to discrete stimuli.

Recent studies utilizing fMRI to study neural response to hunger and satiety states, as well as to food anticipation and ingestion, have mapped discrete areas in the brain which respond to these stimuli. Fuhrer and colleagues found that during hunger, significantly enhanced brain activity is found in the left striate and extrastriate cortex, the inferior parietal lobe, and the orbitofrontal cortices. Stimulation with food images was associated with increased activity in both insulae, the left striate and extrastriate cortex, and the anterior midprefrontal cortex. Nonfood images were associated with enhanced activity in the right parietal lobe and the left and right middle temporal gyrus1. Stice and colleagues reported brain imaging studies which suggested that obese relative to lean individuals show greater activation of the gustatory cortex (insula/frontal operculum) and oral somatosensory regions (parietal operculum and Rolandic operculum) in response to anticipated intake and consumption of palatable foods.

Ghrelin is an orexigenic (appetite stimulating) peptide secreted by the foregut prior to meals and is therefore considered a "meal initiator". Obese patients have low ghrelin levels but maintain a normal diurnal variation of this peptide, while patients after GBP, have reduced ghrelin levels which remain low throughout the day 3. Malik and co-workers demonstrated that when ghrelin was administered intravenously to healthy volunteers during fMRI the neural response to food pictures was affected. The neural effects of ghrelin were correlated with self-rated hunger ratings.

Leptin is an adipocyte-derived circulating hormone that provides information to the brain regarding energy stores. The brain's response to leptin involves changes in energy expenditure and food intake. Farooqi and co-workers reported data suggesting that leptin acts on neural circuits governing food intake to diminish perception of food reward while enhancing the response to satiety signals generated during food consumption.

Peptide YY3-36 (PYY) is a gut-derived satiety signal whose levels increase after meal ingestion. Intravenous infusion of PYY to human volunteers has been shown to cause a decrease in food consumption and self-reported feelings of hunger. It has also been able to alter neuronal activity in within both corticolimbic and higher-cortical areas as well as homeostatic brain regions. Levels of PYY are low in obese subjects, and have has been shown to gradually increase as early as 2 days after GBP, perhaps contributing to the success of this procedure in terms of appetite control.

GLP-1 (glucagons-like peptide 1), like PYY, is an anorexigenic (appetite suppressing) signal. It is secreted from the gut after meals and reduces food intake by an effect on the brain-stem, as well as by decreasing the rate of gastric emptying which adds to the feeling of fullness after a meal. Like PYY, GLP-1 levels are low in obese patients and increase dramatically following GBP, contributing both to the weight loss as well as to the improvement in glucose tolerance after this operation.

Several correlations will be assessed:

1. Correlation between subjective reporting of hunger/satiety and fMRI images.
2. Change in neural response to food-neutral and food-related pictures, following the operation (before vs. 1m and vs. 6m after the procedure).
3. Difference between the two surgical procedures (SG vs.GBP) in regard to the neural response to food images.
4. Correlation between gut-derived appetite-regulating hormone blood levels to subjective reporting of hunger/satiety and fMRI images at the different time points.
5. Correlation of measured parameters to changes in weight, BMI and excess weight loss.

ELIGIBILITY:
Inclusion Criteria:

1. Morbidly obese
2. Having passed standard preoperative, multidisciplinary evaluation and deemed acceptable for surgery

Exclusion Criteria:

1. Claustrophobic
2. Having other cotnraindication for MRI testing (metalic implants, etc.)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-01; Primary Completion 2015-05 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Change in neuronal activity response to visual food stimuli after bariatric surgery | Baseline and 6 months

SECONDARY OUTCOMES:
Change in circulating blood incretin levels after bariatric surgery | Baseline and 6 months
Difference in measured parameters between sleeve gastrectomy and gastric bypass | Baseline and 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel

REFERENCES:
- [Background] Fuhrer D, Zysset S, Stumvoll M. Brain activity in hunger and satiety: an exploratory visually stimulated FMRI study. Obesity (Silver Spring). 2008 May;16(5):945-50. doi: 10.1038/oby.2008.33. Epub 2008 Feb 21. PMID 18292747
- [Background] Stice E, Spoor S, Bohon C, Veldhuizen MG, Small DM. Relation of reward from food intake and anticipated food intake to obesity: a functional magnetic resonance imaging study. J Abnorm Psychol. 2008 Nov;117(4):924-35. doi: 10.1037/a0013600. PMID 19025237
- [Background] Cummings DE, Weigle DS, Frayo RS, Breen PA, Ma MK, Dellinger EP, Purnell JQ. Plasma ghrelin levels after diet-induced weight loss or gastric bypass surgery. N Engl J Med. 2002 May 23;346(21):1623-30. doi: 10.1056/NEJMoa012908. PMID 12023994
- [Background] le Roux CW, Welbourn R, Werling M, Osborne A, Kokkinos A, Laurenius A, Lonroth H, Fandriks L, Ghatei MA, Bloom SR, Olbers T. Gut hormones as mediators of appetite and weight loss after Roux-en-Y gastric bypass. Ann Surg. 2007 Nov;246(5):780-5. doi: 10.1097/SLA.0b013e3180caa3e3. PMID 17968169